CLINICAL TRIAL: NCT07114120
Title: Clinical Study on the Treatment of Stable Bronchiectasis With Bailing Capsules Combined With Guben Kechuan Granules
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: ZhuZhou Central Hospital (Other); Jinhua Central Hospital (Other); Shanghai Zhongshan Hospital (Other); Affiliated Yueqing Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0537
Record Dates: First submitted 2025-06-19; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-06

CONDITIONS: Bronchiectasis; COPD
MeSH Terms: conditions — Bronchiectasis; Pulmonary Disease, Chronic Obstructive | interventions — bailing capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Bailing Capsules orally (four capsules each time, three times a day) and Guben Kechuan Granules (1 bag each time, three times a day) on the basis of standard Western medical treatment
  Interventions: Drug: Bailing Capsules in combination Guben Kechuan Granules
- Control group (No Intervention): standard Western medical treatment

INTERVENTIONS:
Drug: Bailing Capsules in combination Guben Kechuan Granules — Bailing Capsules (four capsules each time, three times a day) in combination Guben Kechuan Granules (1 bag each time，three times a day,)
  Other Names: Bailing Capsules; Guben Kechuan Granules
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to learn if Bailing Capsules in combination Guben Kechuan Granules works to treat stable bronchiectasis in adults.It will also learn about the safety of Bailing Capsules in combination Guben Kechuan Granules The main questions it aims to answer are:

Does Bailing Capsules in combination Guben Kechuan Granules lower the number of acute exacerbation in patients with stable bronchiectasis? The safety of the combination of Bailing Capsules and Guben Kechuan Granules ? Researchers will compare the combination of Bailing Capsules and Guben Kechuan Granules to standard Western medical treatment to see if them works to treat stable bronchiectasis.

Participants will:

Take Bailing Capsules orally (four capsules each time, three times a day) and Guben Kechuan Granules ( three times a day, 1 bag each time )on the basis of standard Western medical treatment or only standard Western medical treatment for 24 weeks Visit the clinic for checkups and tests on 4, 12, 24, 48 weeks Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old, gender not limited;
2. It conforms to the Western medical diagnosis of bronchiectasis;
3. There has been no acute exacerbation or respiratory tract infection in the past 4 weeks. (Acute exacerbation is defined as the deterioration of three or more of the following six conditions: cough, changes in sputum volume, purulent sputum, breathing difficulties or exercise tolerance, fatigue or discomfort, and hemoptysis, lasting for more than 48 hours, and considered by the clinician to require treatment);
4. There have been at least two documented acute exacerbations in the past year, prescribed by doctors and diagnosed as signs and symptoms of respiratory tract infections;
5. Pulmonary function tests can be conducted, and there is evidence of airflow limitation when screening vital capacity (FEV1/FVC ratio <70%, and clinically stable at the time of entering the study);
6. Voluntarily participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Dry bronchiectasis mainly characterized by hemoptysis;
2. Bronchiectasis caused by cystic fibrosis, allergic bronchopulmonary aspergillosis, etc;
3. Previous respiratory diseases other than bronchiectasis (such as bronchial asthma, lung cancer, active pulmonary tuberculosis, interstitial lung disease, pulmonary thromboembolism and severe pneumonia, etc.);
4. Combined with serious diseases of the heart, liver, kidneys, digestive system, blood system, etc., evaluated by the researcher, including but not limited to acute severe hepatitis, liver failure, liver cirrhosis, acute renal failure, acute myocardial infarction, heart failure, gastric perforation, gastrointestinal bleeding, gastric cancer, intestinal cancer, acute leukemia, acute aplastic anemia, etc., subject to the judgment of the researcher;
5. Abnormal liver function was found in the patient screening examination, with the following criteria: total bilirubin > 1.5×ULN; ALT > 3×ULN; AST > 3×ULN;
6. Inability to swallow the research drug;
7. Known allergy to the test drug;
8. Participate in other clinical trials, use other research drugs or research devices within 30 days before randomization;
9. Women or men of childbearing age refused to use contraceptive measures during the study period;
10. Pregnant or lactating women;
11. Any other factors that may not be suitable for participation in clinical research as determined by the researcher;
12. In the past year, there has been a history of alcohol abuse, drug abuse or drug abuse;
13. Other traditional Chinese medicine treatments were used within 7 days before the use of the study drug and during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of acute exacerbations during treatment and follow-up | 24 weeks and 48 weeks

SECONDARY OUTCOMES:
Pulmonary function | 12, 24, 48 weeks
  FVC
Pulmonary function | 12, 24, 48 weeks
  FEV1
Pulmonary function | 12, 24 48 weeks
  FEV1/FVC
Pulmonary function | 12, 24, 48 weeks
  TLC

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - Yueqing People's Hospital, Yueqing, Zhejiang
  - Zhoushan Hospital, Zhoushan, Zhejiang

IPD SHARING:
Plan to Share IPD: No